CLINICAL TRIAL: NCT01942967
Title: Impact of Different Modes of Noninvasive Ventilation (NCPAP Versus TrPA) on Regional Cerebral and Splanchnic Oximetry as Measured by Near Infrared Spectroscopy (NIRS) and Hemodynamics Using Echocardiography in Premature Newborns
Brief Title: Impact of Different Modes of Noninvasive Ventilation on Regional Oximetry and Hemodynamics in Premature Newborn
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Yaser Ali, Fellow, Perinatal-Neonatal Medicine, University of Manitoba
Other Study IDs: B2013: 055
Record Dates: First submitted 2013-07-19; First posted 2013-09-16 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Neonate; Hemodynamic; Tissue oxygenation; Non invasive ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm ≤ 32 weeks GA, on CPAP: Preterm infants less than 32 weeks gestational age requiring CPAP as a mode of respiratory support and admitted in the NICU.While the baby is on CPAP,tissue oxygen saturation monitoring will be started by applying NIRS(Near Infrared Spectroscopy Monitoring) sensors to the forehead and the abdomen. After 3 hours,echocardiography(including Superior Mesenteric Artery Doppler) will be done while the baby is on CPAP. Then, using the same machine, the mode of respiratory support will be changed to TrPA. After another three hours,another echocardiography will be done,then NIRS monitoring will be stopped and the mode of respiratory support will be changed back to CPAP.
  Interventions: Other: Echocardiography; Other: Near Infrared Spectroscopy Monitoring

INTERVENTIONS:
Other: Echocardiography — Measurement of:
  * Left ventricular output (LVO).
  * Right ventricular output (RVO).
  * Assessment of the Mesenteric Artery Flow.
Other: Near Infrared Spectroscopy Monitoring — Measurement of cerebral and mesenteric regional oxygen saturation(rSO2) trends and data while the baby on CPAP or TrPA modes of noninvasive ventilation.
  Other Names: NIRS

SUMMARY:
The purpose of this study is to examine the blood flow and the delivery of oxygen to the brain and gut in preterm babies while they are supported with two modes of breathing machine and compare these two methods to see if one allows for better blood flow to the brain and gut.

DETAILED DESCRIPTION:
Preterm babies under 32 weeks of gestational age usually needs to be supported with breathing machine because of different kinds of problems like lungs immaturity or infection. One type of breathing machine support is called CPAP(Continuous Positive Airway Pressure).This breathing support machine is connected to the nose to help preterm baby breathe. This machine blows air or an air/oxygen mixture through the nose and in to the baby's lung; this helps to keep baby's lungs fully open and makes it easier for the baby to breathe. There are two ways this machine can help the baby breathe - it can either blow the air/oxygen mixture at the same pressure all the time…we call that CPAP, or we can vary the pressure - we call that TrPA(Trigger Pressure Assist). Both methods have been in use in neonatal intensive care units(NICUs) for several years and both methods help with the breathing of babies.

The breathing machine (CPAP) makes the lungs better inflated. This inflation might affect the ability of the heart to push the blood to the organs through the blood vessels. Also we do not know whether there is any difference in the blood flow or oxygen delivery depending whether the baby is on CPAP or TrPA.

We will measure the heart function using Ultrasound (Echocardiography). To measure the efficiency of the flow of the blood through the vessels to the organs we will use Near Infra Red Spectroscopy (NIRS); this involves applying a sensor to the baby's skin - one on the forehead and one on the tummy and connecting the sensors to a machine which can measure the oxygen level in the organ under the skin.

While the baby is on CPAP, we will start monitoring oxygen saturation by applying NIRS sensors to the forehead and the abdomen. After 3 hours we will do echocardiography (ultrasound of the heart)to see any changes that might happen to the heart and blood vessels while the baby is on CPAP. Then, using the same machine, we will change the mode of respiratory support to TrPA. After another three hours, we will do another echocardiography (ultrasound of the heart), then we will stop NIRS monitoring and change the mode of respiratory support back to CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 34 weeks gestational age
* Requirement of CPAP or TrPA as a mode of respiratory support

Exclusion Criteria:

* Lack of parental consent
* Preterm infants more than 34 gestational weeks
* Preterm infants with congenital malformation
* Severe perinatal asphyxia
* Hemodynamically significant patent ductus arteriosus (PDA)
* Pulmonary hypertension
* Septic shock
* Any associated congenital heart diseases other than non-significant PDA or patent foramen ovale (PFO)
* Stage 2 or 3 necrotising enterocolitis (NEC)
* Intraventricular hemorrhage (IVH) grade 3 or 4

Ages: 48 Hours to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants less than 34 weeks gestational age at birth Requiring CPAP or TrPA as a mode of respiratory support
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output | Day 3 of life till 2 months of age
  Targeted neonatal Echocardiography will be done according to the guidelines accepted by the writing group of the American society of echocardiography in collaboration with associations of European pediatric cardiologists
  The following standard windows will be used:
  1. Subcostal.
  2. Apical.
  3. Long and short axis parasternal.
  4. Suprasternal
  Measurements:
  * Left ventricular output (LVO).
  * Right ventricular output (RVO).
Changes in Superior Mesenteric Artery and Middle Cerebral Artery Doppler flow. | Day 3 of life till 2 months of age
Cerebral and mesenteric regional tissue oxygenation | Day 3 of life till 2 months of age
  Cerebral and mesenteric rSO2 trends and data (obtained by NIRS) will be recorded along with simultaneous pulse oximeter trends and data. The splanchnic-cerebral oxygenation ratio (SCOR) reflecting the ratio between regional cerebral oxygen saturation(rcSO2) and regional splanchnic oxygen saturation (rsSO2)(rcSO2/rsSO2) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Srinivasan, MD, Study Director — University of Manitoba; Mary S Seshia, MD, Study Director — University of Manitoba
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Center, Winnipeg, Manitoba